CLINICAL TRIAL: NCT05819385
Title: Ambispective, Non-Interventional Study to Evaluate the Epidemiology of Interstitial Lung Diseases (ILDs) Associated to Rheumatic Diseases (Rheumatoid Arthritis, Connective Tissue Diseases, Spondylarthritis and Sarcoidosis) and the Progression Risk Factors in the Mexican Population
Brief Title: Connective Tissue Disease-associated Interstitial Lung Diseases (CTD-ILD) Epidemiology Non-interventional Study (NIS)
Status: Recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: TIC Social Mexico (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1199-0522
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All participants must be diagnosed with rheumatic disease (connective tissue disease (CTD)) and intestinal lung disease (ILD) and fulfil all inclusion and no exclusion criteria. Information about participants will be obtained from electronic and physical medical records for existing data collection (over the past ten years, from 2012 to 2022) and/or from medical consultations for newly collected data (for the next three years, from 2023 to 2026). The participants' observation time varies and can be over the whole study duration (from 2012 to 2023), over the past ten years only (existing data) or over the next three years (new data).

SUMMARY:
This study aims to characterize the epidemiology of interstitial lung diseases (ILD) associated to connective tissue disease (CTD) in Mexico, and to study its correlation with the different comorbidities and treatments used, as well as the possible impacts of these factors on the outcome of progression, exacerbations, and mortality in patients with ILD associated to CTD.

ELIGIBILITY:
Inclusion Criteria:

For newly data collection:

* Male and female Patients.
* Patients over 18 years old.
* Patient who gives his/her signed informed consent to be able to use information about their condition.
* Patient who has the diagnosis of: rheumatoid arthritis, connective tissue disease (CTD) (systemic sclerosis or scleroderma; inflammatory myopathy: antisynthetase, dermatomyositis, polymyositis, mixed connective tissue disease; systemic lupus erythematosus; primary Sjögren syndrome; pulmonary fibrosis associated with non-specific autoimmunity; primary systemic vasculitis; psoriasis, anchylosing spondylitis, reactive arthritis) Spondyloarthritis (SpA) or sarcoidosis, (accordingly with the updated clinical criteria for each pathology).

Patient with any interstitial lung diseases (ILD) diagnosed clinically and by a high-resolution computed tomography study with an interstitial pattern (supervised by an expert radiologist).

For existing data collection:

* Medical Records from patients with whom contact was permanently lost for any reason since 2012 till the study start date.
* Medical Records from male and female Patients.
* Medical Records from patients over 18 years old.
* Medical Records of patients that have at least: patient initials, date of birth, gender, date of diagnosis, full diagnosis of:

  * Patient who has the diagnosis of: rheumatoid arthritis, CTD (systemic sclerosis or scleroderma; inflammatory myopathy: antisynthetase, dermatomyositis, polymyositis, mixed connective tissue disease; Systemic lupus erythematosus; primary Sjögren syndrome; pulmonary fibrosis associated with non-specific autoimmunity; primary systemic vasculitis; psoriasis, anchylosing spondylitis, reactive arthritis) SpA or Sarcoidosis, (accordingly with the updated clinical criteria for each pathology).
  * Patient with any ILD diagnosed clinically and by a high-resolution computed tomography study with an interstitial pattern (supervised by an expert radiologist).

Exclusion Criteria:

* Patient with a biopsy definition of usual interstitial pneumonitis, related to any other non-CTD.
* Patient with post-chemotherapy or post-radiotherapy pneumonitis.
* Medical Records of patients without full diagnostic of ILD (clinically and by biopsy or high-resolution computed tomography).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants must be diagnosed with rheumatic disease (connective tissue disease (CTD)) and intestinal lung disease (ILD) and fulfil all inclusion and no exclusion criteria. Information about participants will be obtained from electronic and physical medical records for existing data collection (over the past ten years, from 2012 to 2022) and/or from medical consultations for newly collected data (for the next three years, from 2023 to 2026). The participants' observation time varies and can be over the whole study duration (from 2012 to 2023), over the past ten years only (existing data) or over the next three years (new data).
Sampling Method: Probability Sample
Enrollment: 312 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to first exacerbation: time in months elapsed until the first exacerbation from the diagnosis | up to 13 years
Number of exacerbation per year (frequency of exacerbation) | up to 13 years
Percent of pulmonary fibrosis: grade of parenchymal involvement evidenced by high-resolution computed tomography (HRCT) | up to 13 years
Change in 6-minute walk tests (6-MWT) over time | up to 13 years
King's Brief Interstitial Lung Disease Questionnaire (K-BILD) score change over time | up to 13 years
Saint George Respiratory Questionnaire (SGRQ)-I score change over time | up to 13 years

SECONDARY OUTCOMES:
Possibility to have an exacerbation and/or progression in pulmonary fibrosis, sorted by rheumatic disease type (rheumatoid arthritis (RA), connective tissue disease (CTD), spondyloarthritis (SpA) and Sarcoidosis) | up to 13 years
Frequency of use of diagnostic tools (laboratory, cabinet) | up to 13 years
Progression of pulmonary fibrosis by treatment received identified by HRCT patterns, lung function, activity score and damage index | up to 13 years

CONTACTS AND LOCATIONS:
Locations (1):
- Colegio Mexicano de Reumatología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Once the criteria in section 'time frame frame' are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com